CLINICAL TRIAL: NCT00003119
Title: Primary Surgical Therapy for Biologically Defined Low-Risk Neuroblastoma: A Pediatric Oncology Group/Children's Cancer Group Intergroup Study
Brief Title: Surgery in Treating Children With Neuroblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P9641; COG-P9641 (Other: Children's Oncology Group); POG-P9641 (Other: Pediatric Oncology Group); CCG-P9641 (Other: Children's Cancer Group); CDR0000065874 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Neuroblastoma
Keywords: localized resectable neuroblastoma; stage 4S neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; sargramostim; Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment 1 - Asymptomatic - no immediate chemotherapy (Experimental)
  Interventions: Procedure: conventional surgery; Radiation: radiation therapy
- Symptomatic - immediate chemotherapy (Experimental)
  Interventions: Biological: filgrastim; Biological: sargramostim; Drug: carboplatin; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Procedure: adjuvant therapy; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
  Arms: Symptomatic - immediate chemotherapy
Biological: sargramostim
  Arms: Symptomatic - immediate chemotherapy
Drug: carboplatin
  Arms: Symptomatic - immediate chemotherapy
Drug: cyclophosphamide
  Arms: Symptomatic - immediate chemotherapy
Drug: doxorubicin hydrochloride
  Arms: Symptomatic - immediate chemotherapy
Drug: etoposide
  Arms: Symptomatic - immediate chemotherapy
Procedure: adjuvant therapy
  Arms: Symptomatic - immediate chemotherapy
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Surgery alone may be effective in treating children with neuroblastoma.

PURPOSE: Phase III trial to study the effectiveness of surgery alone in treating children who have neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if asymptomatic patients with low-risk neuroblastoma treated with surgery alone will have a 3-year survival rate of 95%.
* Estimate the response and 3-year event-free survival rates of symptomatic patients treated with chemotherapy.
* Estimate the event-free survival and overall survival rates in patients who relapse or progress after initial treatment with surgery alone.
* Determine the acute and chronic toxic effects associated with treating low-risk neuroblastoma with surgery alone or surgery and chemotherapy.

OUTLINE: This is a multicenter study. Patients are stratified according to disease stage, MYCN status, age, and histology.

Patients undergo primary tumor resection and biopsy of regional nodes. Patients with at least 50% of the tumor resected are followed monthly for 3 months, every 3 months for 9 months, every 6 months for one year, and then annually thereafter.

Regimen I

* Patients with clinically symptomatic (e.g., respiratory distress, spinal cord compromise with or without neurologic deficit, inferior vena cava compression with renal or bowel ischemia, intractable vomiting due to gastrointestinal obstruction, genitourinary obstruction, or coagulopathy) low-risk neuroblastoma or who have less than 50% of the primary tumor resected receive 4 different courses of chemotherapy.
* Course 1: Patients receive carboplatin IV over 1 hour followed by etoposide IV over 2 hours on day 0 and etoposide only on days 1 and 2.
* Course 2: Patients receive carboplatin IV over 1 hour, cyclophosphamide IV over 1 hour, and doxorubicin IV over 15-60 minutes on day 1.
* Course 3: Patients receive cyclophosphamide IV over 1 hour followed by etoposide IV over 2 hours on day 0 and etoposide only on days 1 and 2.
* Course 4: Patients receive carboplatin IV over 1 hour and etoposide IV over 2 hours followed by doxorubicin IV over 15-60 minutes on day 0 and etoposide only on days 1 and 2.

Regimen II

* Patients who progress to or recur with unfavorable biology intermediate-risk disease receive an additional 4 courses of chemotherapy.
* Course 5: Patients receive treatment as in course 3 above.
* Course 6: Patients receive treatment as in course 2 above.
* Course 7: Patients receive treatment as in course 1 above.
* Course 8: Patients receive cyclophosphamide IV over 1 hour followed by doxorubicin IV over 15-60 minutes on day 1.

All infants under 60 days of age receive filgrastim (G-CSF) or sargramostim (GM-CSF) subcutaneously beginning 24 to 36 hours after chemotherapy and continuing until blood counts recover.

Courses in both regimens repeat every 3 weeks in the absence of unacceptable toxicity.

Patients at risk for symptomatic spinal cord compression may also receive chemotherapy. Patients experiencing progressive or recurrent disease after observation undergo repeat surgery and/or chemotherapy as above. Patients with clinically symptomatic disease may also undergo radiotherapy if response to chemotherapy is not rapid.

Patients are followed every 2 months for 1 year, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 820 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven low-risk neuroblastoma (excluding ganglioneuroma)

  * International Neuroblastoma Staging System (INSS) stage 1 in all patients
  * INSS stage 2A or 2B in patients less than 365 days of age
  * INSS stage 2A or 2B tumor with nonamplified MYCN with any Shimada histology in patients ages 1 to 20 years
  * INSS stage 2A or 2B tumor with amplified MYCN with Shimada favorable histology in patients ages 1 to 20 years
  * INSS stage 4S tumors with nonamplified MYCN, Shimada favorable histology, and a DNA index not equal to 1 in patients less than 365 days of age
* Immediate chemotherapy allowed prior to biopsy for patients with intradural extension and/or emergent paresis if biopsy performed within 96 hours

  * Must have no abnormal organ function unless due to neuroblastoma
* Concurrent registration on companion biology study (protocol COG-ANBL00B1) or its successor

PATIENT CHARACTERISTICS:

Age:

* Under 21

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 1.5 times normal
* SGOT or SGPT less than 2.5 times normal

Renal:

* Creatinine less than 1.5 times normal

Cardiovascular:

* Shortening fraction greater than 27% by echocardiogram OR
* Ejection fraction greater than 47% by radionuclide angiogram

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* No prior hormonal therapy

Radiotherapy:

* No prior radiotherapy

Surgery:

* Prior surgery allowed

Other:

* No other prior therapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 968 (Actual)
Dates: Start 1998-03; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Estimate the 3 year survival rate for low risk asymptomatic stage 2A/2B patients who are treated with surgery alone
  The primary objective is to estimate the 3 year survival rate for low risk asymptomatic stage 2A/2B patients who are treated with surgery alone. Under the assumption that about 90% of the low risk 2A/2B patients will be asymptomatic, and 10% of these will be lost to follow up, the projected sample size will enable estimation of the survival rate with a standard error less than .03. This sample size will also provide sufficient power for the sequential monitoring plan (see below) for this subgroup of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R. Strother, MD, Study Chair — Alberta Children's Hospital
Locations (235):
- United States (207):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Cancer Research Institute, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital and Health Center, San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - University of Connecticut Comprehensive Cancer Center at University of Connecticut Health Center, Farmington, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Mountain States Tumor Institute - Boise, Boise, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Medical Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - St. Vincent Hospitals and Health Care Centers, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Walter Reed Army Medical Center, Silver Spring, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Baystate Regional Cancer Program at Baystate Medical Center, Springfield, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health and DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Hospitals and Clinics - Minnesota, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Valerie Fund Children's Center at Atlantic Health, Summit, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Comprehensive Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center of University Health Systems of Eastern Carolina, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Dakota Cancer Institute at Innovis Health - Dakota Clinic, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Forum Health-Tod Childrens Hospital, Youngstown, Ohio
  - Children's Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Doernbecher Children's Hospital at Oregon Health & Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital at University of South Dakota Medical Center, Sioux Falls, South Dakota
  - East Tennessee State University Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas
  - Methodist Cancer Center at Methodist Specialty and Transplant Hospital, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Center for Cancer Prevention and Care at Scott and White Clinic, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Carilion Medical Center for Children, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Cabell Huntington Hospital, Huntington, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (6):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier de l'Universite Laval, Sainte-Foy, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- Starship Children's Health, Auckland, New Zealand
- Puerto Rico (2):
  - Puerto Rico Cancer Center at University of Puerto Rico - Medical Sciences Campus, San Juan
  - San Jorge Childrens Hospital, Santurce
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Background] Meany HJ, Attiyeh EF, Naranjo A, et al.: Outcome analysis of non-high-risk neuroblastoma patients enrolled on Children's Oncology Group trials P9641 and A3961. [Abstract] J Clin Oncol 30 (Suppl 15): A-9533, 2012.
- [Background] Attiyeh EF, Mosse YP, Diskin S, et al.: Identification of genomic DNA signatures predicting relapse in low- and intermediate- risk neuroblastoma using a case control design and high-density SNP genotyping: a Children's Oncology Group (COG) study. [Abstract] J Clin Oncol 25 (Suppl 18): A-9500, 526s, 2007.
- [Result] Strother DR, London WB, Schmidt ML, Brodeur GM, Shimada H, Thorner P, Collins MH, Tagge E, Adkins S, Reynolds CP, Murray K, Lavey RS, Matthay KK, Castleberry R, Maris JM, Cohn SL. Outcome after surgery alone or with restricted use of chemotherapy for patients with low-risk neuroblastoma: results of Children's Oncology Group study P9641. J Clin Oncol. 2012 May 20;30(15):1842-8. doi: 10.1200/JCO.2011.37.9990. Epub 2012 Apr 23. PMID 22529259